CLINICAL TRIAL: NCT03309124
Title: Effect of White Potatoes on Glycemic Response and Satiety in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB2017-330
Record Dates: First submitted 2017-09-29; First posted 2017-10-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: White potatoes; Older adults; Satiety; Glycaemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- White bread (Experimental): Matched for energy content and available carbohydrate content of potato treatments
  Interventions: Other: White bread
- Baked potato with skin (Experimental): Baked russet potato
  Interventions: Other: Baked potato with skin
- Mashed potatoes (Experimental): Mashed potatoes prepared from frozen, matched for available carbohydrate content of baked potato
  Interventions: Other: Mashed potatoes
- Fried French fries (Experimental): Matched for available carbohydrate content of baked potato
  Interventions: Other: Fried French fries
- Meal skipping (Experimental): No food given
  Interventions: Other: Meal skipping

INTERVENTIONS:
Other: White bread — Toasted, with canola oil added to match for fat content of French fries (13.9 grams), as well as being matched for energy (280 kilocalories) and available carbohydrate content (33 grams) of potato treatments.
  Arms: White bread
Other: Baked potato with skin — Baked russet potato with canola oil added once baked to match for fat content of French fries, and also matched for the salt content of white bread (280 milligrams).
  Arms: Baked potato with skin
Other: Mashed potatoes — Mashed potatoes prepared from frozen, with canola oil added to match for fat content of French fries, as well as being matched for energy and available carbohydrate content of the baked potato.
  Arms: Mashed potatoes
Other: Fried French fries — Prepared from frozen, matched for energy and available carbohydrate content of baked potato and salt content of white bread.
  Arms: Fried French fries
Other: Meal skipping — No food given
  Arms: Meal skipping

SUMMARY:
The purpose of the present study is to explore the influence of cooking methods of potatoes on post-prandial glycaemia and satiety in healthy older adults.

DETAILED DESCRIPTION:
Each of the 5 study sessions will be at least 7 days apart. Either meal skipping, or one of three treatments of white potatoes (a) baked (with skin), (b) mashed, (c) fried French fries, or white bread, prepared on the day of testing, will be served to healthy older adults (65+ years). Participants will consume the equivalent to 1 medium sized potato (~280 kcal) or an equivalent amount of calories from white bread. Glycemic response, insulin, incretin hormones (glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic peptide (GIP)), dipeptidyl peptidase 4 (DPP4), and cholecystokinin (CCK) will be measured for 2 h (0, 15, 30, 45, 60, 90 and 120 min) following meal consumption, as well as mood and subjective appetite. An ad libitum test meal will be provided at 120 min to assess food intake suppression.

ELIGIBILITY:
Inclusion Criteria:

* be 65 years or older
* be healthy
* not be taking medications that affect food intake regulation or blood glucose

Exclusion Criteria:

* anyone with food sensitivities or allergies to potatoes or potato-products,
* smokers
* diabetic or overweight/obese individuals.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake (lunch, at 120 minutes) | 120 minutes after meal consumption
  Food intake will be determined by weighing the meal before and after serving. The net weight of the test meal will be converted to calories
Change from baseline glycemic response | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Blood glucose (mmol/L). Blood glucose will be measured in whole blood using YSI 2300 STAT PLUS (YSI Incorporated, Yellow Springs, OH)
Change from baseline insulin | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Blood insulin (pmol/L). Insulin concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).

SECONDARY OUTCOMES:
Change from baseline subjective appetite | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Measured using visual analogue scale (mm). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings.
Change from baseline mood | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Measured using visual analogue scale (mm). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings.
Change from baseline cholecystokinin (CCK) | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Blood CCK (pmol/L). CCK concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts)
Change from baseline dipeptidyl peptidase 4 (DPP4) | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Blood DPP4 (ng/mL). DPP4 concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts)
Change from baseline glucose-dependent insulinotropic peptide (GIP) | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Blood GIP (pmol/L). GIP concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts)
Change from baseline glucagon-like peptide-1 (GLP-1) | baseline and then 15, 30, 45, 60, 90 and 120 minutes after meal consumption
  Blood GLP-1 (pmol/L). GLP-1 concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided